CLINICAL TRIAL: NCT05158556
Title: Gender Based Comparison of Myofascial Release Technique and Instrument Assisted Soft Tissue Mobilization on Trigger Points in Lumbar Region
Brief Title: Comparison of Myofascial Release Technique and Instrument Assisted Soft Tissue Mobilization in Lumbar Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-00936 Irum Nosheen
Record Dates: First submitted 2021-12-13; First posted 2021-12-15 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: trigger point,; myofascial release; instrument assisted soft tissue mobilization; range of motion; pain
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- myofascial release technique (Experimental): Myofascial Release Technique will be applied with forearm/ ulnar border of palm. deep pressure will be applied and glided medially towards the thoraco-lumbar region.ins
  Interventions: Other: Myofascial Release Technique; Other: Instrument Assisted Soft tissue Mobilization
- Instrument Assisted Soft Tissue Mobilization (Experimental): instrument assisted soft tissue mobilization is done via M2T Blade. it is a multifunctional instrument consisting of many planes and is very effective in treating pain and spasm. Its efficacy is proven over soft tissues that it releases fascial tightness.
  Interventions: Other: Myofascial Release Technique; Other: Instrument Assisted Soft tissue Mobilization

INTERVENTIONS:
Other: Myofascial Release Technique — Myofascial Release Technique will be applied with forearm/ ulnar border of palm. Deep pressure will be applied and glided medially towards the thoraco-lumbar region.
Other: Instrument Assisted Soft tissue Mobilization — instrument assisted soft tissue mobilization is done via M2T Blade. it is a multifunctional instrument consisting of many planes and is very effective in treating pain and spasm. Its efficacy is proven over soft tissues that it releases fascial tightness.

SUMMARY:
Trigger point are hyper-irritable points, appear as nodules on palpation, discrete and focal spots in the taut band of skeletal muscles. Myofascial release technique and instrument assisted soft tissue mobilization both techniques are used to break the adhesions and mobilize the soft tissue, releasing the trigger points. The study will contribute in comparing the level of pain threshold perceived by males and females in our society. .Moreover, finding a noninvasive effective treatment that is non-exhaustive for the therapist and non-painful for the patient.

DETAILED DESCRIPTION:
Trigger points are hyper-irritable points, appear as nodules on palpation, discrete and focal spots in the taut band of skeletal muscles. Usually these points are sensitive to pressure, if direct compression is applied over them, that can evoke jump sign, tenderness and pain is produced locally but it is referred to surrounding areas. There are many types of trigger points on the basis of location, chronicity and tenderness. They are classified as central, satellite, diffuse, inactive,and active. The trigger points can be developed by repetitive overuse injuries or sustained loading like lifting heavy weight, carrying babies, bags, briefcase etc. It can also be manifested by poor posture or prolonged period of inactivity such as bed rest or sitting causing pain, reduced range of motion, muscle tightness. When there are number of trigger points in muscles causing micro-cramps resulting in myofascial pain syndrome. Trigger points are the areas of contracted muscles causing restriction of in blood flow within the tissues. She claimed that by applying sustained pressure over trigger points with thumbs, knuckles and elbow followed by stretching of the muscle produced much better results compared to trigger point injections. Myofascial trigger points in lumbar region play an important role in genesis of mechanical low back pain. The hyper-irritable spots usually present within the taut band of skeletal muscles which on compression can give rise to characteristics like; referred pain, autonomic phenomena like (sweating, vasoconstriction and pilomotor activity) and motor dysfunction. It is essential to inquire the gender differences in pain perception level because many diseases like migraine, rheumatoid arthritis, and low back pain are more common among females than males. Females not only report more pain but they also experience more intense pain in their body parts as compared to males. Factors like psychological and physiological contribute in difference in pain perception among females and male. A study suggests that females show greater perception towards pain threshold as compared to males.

Myofascial release technique is usually considered as alternative of medicine therapy highly recommended to treat immobility of skeletal muscles and pain by improving blood circulation and oxygen in these muscles and is non-invasive method. Moreover, it produces stretch reflex in muscles. By applying sustained pressure for 30 seconds over the trigger points until the patient's pain intensity is decreased considerably. As this pressure applied would help to break the adhesive fibres connection within the muscle helping to push out the blood containing waste products and toxins because after 30 seconds fresh blood containing nutrients will flow and trigger points are released.

Instrument assisted soft tissue mobilization (IASTM) is also a professional practice to treat soft tissues. Moreover, IASTM mainly decreases pain sensitivity and pain threshold of myofascial trigger points. It is applied by using the instrument made up of stainless steel with edges and contours according to different body locations allowing deeper penetration treating soft tissue disorders. Instrument assisted soft tissue mobilization is master intervention using specialized tool to manipulate the skin , muscles, myofascial, tendons by various direct compressive strokes. IASTM technique is very effective as it effectively break the restrictions in fascia and scar tissue. Adhesions may developed within the soft tissue after surgery, immobilization, strain, are broken down by using this instrument allowing full restoration of function.

The tool I am using in my study for instrument assisted soft tissue mobilization technique is M2T Blade technique is a multifunctional instrument invented by Adam Broger consisting of many planes and is very effective in treating pain and spasm. M2T Blade is a new invention and it is beneficial in reducing myofascial pain. Its efficacy is proven over soft tissues that it releases fascial tightness. Moreover it also improves range of motion of a joint. Highly loaded blades are designed to provide a specific distribution is given. The three-dimensional analysis methodology is used here.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one active trigger point in lumbar region.
* Office workers sitting in office > 5 hours a day.
* Targeting both deep and superficial muscles.

Exclusion Criteria:

* History of spinal surgeries
* Trauma
* Acute Fractures
* Tuberculosis spine
* Wounds, Infections or any other cause of back pain.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | for 6 weeks
  Numeric Pain Rating Scale is an 11 point tool used to assess the pain intensity among people. Its value ranges from 0 to 10, where 0 means no pain and 10 means worst possible pain. It is a reliable and valid tool (r=0.96, its validity correlations range from 0.86 to 0.95.Assesment was performed at the base line and after 6-weeks.
Pain Sensitivity Questionnaire | for 6 weeks
  Pain sensitivity questionnaire is a valid and reliable tool used to measure pain perception in different populations. Cronbach's alpha value for the Pain Sensitivity Questionnaire was 0.92. Assesment was performed at the base line and after 6-weeks.
inclinometer | for 6 weeks
  An inclinometer is a device used by physical therapist to measure range of motion for spinal posture. An inclinometer gives more accurate, precise and reproducible Range of motion measurements than goniometer. It is a reliable and valid tool r=0.93, validity=0.92. Assesment was performed at the base line and after 6-weeks.
Modified Somatic Perception Questionnaire | for 6 weeks
  Modified Somatic Perception Questionnaire is a self-report scale consists of 13 items. It helps to find out the complaints that are associated with psychological responses. The scale has ICC value 0.72. Assesment was performed at the base line and after 6-weeks.
algometer | for 6 weeks
  Algometer is a reliable and valid tool used to measure the pressure pain threshold. intraclass correlation coefficient value =0.91. Assesment was performed at the base line and after 6-weeks.

CONTACTS AND LOCATIONS:
Overall Officials: maria khalid, Ms-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Muzaffar Khan Surgical Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No